CLINICAL TRIAL: NCT00561535
Title: Effect of a Probiotic, Lactobacillus FARCIMINIS, in Diarrhea Predominant IBS
Brief Title: Effect of a Probiotic, Lactobacillus FARCIMINIS, in Diarrhea Predominant IBS Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Association pour l'Etude des Fonctions Digestives (Unknown)
Responsible Party: COFFIN, Association pour l'Etude des Fonctions Digestives
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AEFD 2007-01
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2011-01

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS; Diarrhea; Rome III
MeSH Terms: conditions — Irritable Bowel Syndrome; Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Lactobacillus FARCIMINIS
  Interventions: Dietary Supplement: Lactobacillus FARCIMINIS
- B (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: placebo (starch)

INTERVENTIONS:
Dietary Supplement: Lactobacillus FARCIMINIS — 10.10 UFC of lactobacillus FARCIMINIS
  Other Names: 10.10 UFC of lactobacillus FARCIMINIS
  Arms: A
Dietary Supplement: placebo (starch) — Once daily
  Other Names: Once daily
  Arms: B

SUMMARY:
Probiotics may improve symptoms in IBS patients. The aim of this study is to test the efficacy of Lactobacillus FARCIMINIS in diarrhea predominant IBS patients according to Rome III criteria.

DETAILED DESCRIPTION:
The aim of this study is to test the efficacy of Lactobacillus FARCIMINIS in diarrhea predominant IBS patients according to Rome III criteria.

ELIGIBILITY:
Inclusion Criteria:

* Diarrhea predominant IBS
* Less than 5-year duration
* Pain intensity between 2 and 7 on VAS

Exclusion Criteria:

* Celiac disease
* Antibiotic treatment within the 1-month period preceding inclusion
* Digestive organic disease
* Any severe non digestive organic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-10; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Overall subject's assessment | 4 weeks

SECONDARY OUTCOMES:
Decrease in abdominal pain, stool form and consistency, modifications in intestinal permeability, modification in fecal serine protease activity, modifications in interleukin seric concentrations | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Coffin, Prof, Principal Investigator — Assistance Publique Hopitaux de Paris; Yoram Bouhnik, Prof, Study Director — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Louis Mourier, GI Unit, Colombes, Île-de-France Region, France

REFERENCES:
- [Background] Camilleri M, Chang L. Challenges to the therapeutic pipeline for irritable bowel syndrome: end points and regulatory hurdles. Gastroenterology. 2008 Dec;135(6):1877-91. doi: 10.1053/j.gastro.2008.09.005. Epub 2008 Oct 9. PMID 18848833